CLINICAL TRIAL: NCT06717620
Title: Influcence Oj Stress on Body Composition During Exam Preparation
Brief Title: Changes in Body Composition During Exam Period
Status: Completed | Type: Observational
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Natalia Mudarra García, Doctor in health care. Principal Investigator. Clinical Professor, Universidad Complutense de Madrid
Other Study IDs: ACT 244.23. Puerta de Hierro
Record Dates: First submitted 2024-11-13; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Body Weight Changes
Keywords: Diet Healthy; Body Composition; Exercise; Stress Psychological
MeSH Terms: conditions — Body Weight Changes; Motor Activity; Stress, Psychological

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- UCM students: Measurements before and after the exam period
  Interventions: Behavioral: Body composition before and after exams

INTERVENTIONS:
Behavioral: Body composition before and after exams — Measurement of body composition, eating habits, physical exercise in the same group of students before and after the exams

SUMMARY:
Introduction: Academic stress is defined as an activation reaction to stimuli and academic events that can cause alterations in diet and physical exercise. Students are the population most at risk of leading an unhealthy life as a result of stress. These bad habits and leading a sedentary lifestyle can cause an alteration in body composition and increase the risk of diseases.

Methodology: This is an observational, comparative, prospective and longitudinal study based on the collection of data from the same group of students at two different stages of the year (before exam preparation, January 2024 and during exam preparation, May 2024).

The tests carried out to assess eating habits, physical exercise and body composition were the Kidmed survey, the IPAQ test and measurement with a bioimpedance meter, respectively.

DETAILED DESCRIPTION:
INTRODUCTION:

Thanks to good eating habits, people can lead a healthy life. All these habits are related to the way in which people select a food, process it and consume it, since it must provide our body with the necessary nutrients so that it is later able to perform vital functions. To have a healthy diet it depends on a series of factors such as food processing, eating time and stress and anxiety. Eating a healthy diet helps to prevent diseases such as hypertension, cancer, anemia, obesity and osteoporosis.

Young people from their childhood acquire a series of habits that they build throughout their lives according to the style they have, being influenced by their culture, customs and beliefs, among others. All this can generate food tastes and certain behaviors that can favor or harm true healthy practices. Nowadays, the population is consuming more and more fast food (ultra-processed foods, high in fat and sugar) and is increasingly sedentary, since it occupies most of its free time in activities that include the use of screens, video consoles and mobile phones. This sedentary lifestyle causes negative consequences, both physical and social. A healthy diet always has to be linked to exercise. It should be done daily, avoiding physical inactivity and a sedentary lifestyle.

Physical exercise plays a very important role in the body. As the amount of physical exercise we do increases, our respiratory system improves lung capacity and we are less likely to contract respiratory diseases. Physical exercise also improves mental hygiene, (it helps us to reduce that stress or anxiety we suffer), so it is essential to do sports when students have exams as this will help them to increase our level of concentration.

Stress is a short-term response of the human body to a threatening situation. When it appears, it causes alterations in diet and physical exercise. We can find two manifestations of stress: organic and psychological. In the latter, there is academic stress, which is the focus of this research. It is defined as a physiological, emotional, cognitive, and behavioral activation reaction to stimuli and academic events. Students are the population most at risk of leading an unhealthy life because they undergo numerous exams every year that in one way or another cause them stress. Most of the time this stress is a consequence of competitiveness (competing to be better) of the objectives set by the student (getting a job as soon as possible, being able to opt for the desired university career, managing time well to be able to prepare many subjects at the same time, etc.).or because of the unachieved objectives that frustration entails. This stress can also be increased by an overload of work, since they not only have to study for exams, but also have to go to practices, talks or do work in each subject. All this increased stress can be detrimental in the future.

Body composition is a concept that refers to the main components that constitute the human body, these are: bone, water, muscle, fat and visceral tissue (A visceral tissue greater than 12% indicates that upper abdominal fat is beginning to infiltrate, which is quite dangerous for our nutritional health, since if it is not corrected it can indicate more predisposition to cardiovascular and metabolic diseases). These components can be measured by a bioimpedance meter, whose operation consists of an electrical impulse that runs between two poles of the body as if from hand to hand, or from foot to foot (which is why it is necessary for the person to take off their shoes) calculating the time it takes for this impulse to travel that distance. In this way, the amount and percentage of each of these elements can be estimated. Eating an unhealthy diet and a more sedentary life leads to many alterations in body composition.

As we well know, students are subjected to high periods of stress, especially during exam time, due to the above. All this stress means that they develop bad habits, such as making changes in their diet (eating unhealthy foods, or eating excess or insufficient amounts) and alterations in their sports routines (since due to lack of time they cannot do the same sport as before), which could cause an alteration in body composition and increase the risk of diseases.

The purpose of this study is to demonstrate how stress and anxiety to which students are subjected during the exam period leads to a change in body composition, due to poor diet and lack of physical exercise. With the results obtained, improvements can be implemented and young people can be made aware of the importance of healthy habits.

The main objective was to evaluate the body composition of university students by relating the food they ate and the physical exercise they performed before and during the exam period.

METHODOLOGY Design, population, sample

This is an observational, prospective, comparative, prospective and longitudinal study carried out on students of the Faculty of Nursing of the Complutense University of Madrid. To calculate the sample size, a 15% loss, a confidence level of 95%, an accuracy of 3% and a proportion of 5% were assumed. An adequate sample size of 140 was estimated. A convenience sampling was carried out.

Students over 18 years of age, students enrolled in the second year of the Bachelor's Degree in Nursing, students belonging to the Complutense University of Madrid were included. The students who were excluded from the study had some physical inability to perform impedancemetry, were not going to take the exam of the subject or were on pharmacological treatments such as thyroid hormones etc...

Study variables

The following sociodemographic and clinical variables were collected: age, sex (female, male), weight, height, ethnicity (Asian, European, American, African), body composition was measured by bioimpedance meter (Suplementary info III) BEURER BF 1000 (muscle mass, fat mass, visceral tissue), eating habits were measured with the modified KIDMED questionnaire (Suplementary table I), physical exercise performance using the IPAQ international physical exercise questionnaire (Supplementary table II), Smoke (yes and no), drink caffeine (yes and no), drink Coca Cola (yes and no), take stimulant drugs (yes and no).

Intervention Once the students agreed to enter the study, they were given the kidmed I survey (12) to evaluate eating habits, the IPAQ physical exercise survey (13) to calculate the physical exercise they performed, and the bioimpedance meter (BEURER BF 1000 brand) to calculate body composition.

This data collection was carried out in two stages of the year. The first data extraction was before the examination period (January 2024), where the parameters described above (sociodemographic variables, bioimpedancemetrics, eating habits and physical exercise) were collected.

The second part of the research was carried out after the end of the examination stage (last week of May 2024). At this time, body composition was assessed again and they were given the diet and physical exercise survey to answer the questions, focused on the habits they had carried out the 7 days before the exams. After data collection, the data collected on body composition were compared with eating and physical exercise habits.

Finally, the results collected in the first stage were compared with the data collected in the second, only from the students who had taken both (since some did not attend the second assessment), to see if the stress caused by the exams influenced lifestyle habits such as diet and physical exercise and the morphofunctional assessment (assessment of fat mass, muscle mass and visceral tissue).

All data were collected in a database (REDCAP) specially designed for this study by the researchers (N.M., F.G., M.P., I.O. and MJ.V.).

This study was approved by the Ethics and Research Committee of the Puerta de Hierro University Hospital (ACT 244/23). Access to the study files has been password protected and restricted to the responsible researchers (N.M., F.G., M.P., I.O. and MJ.V.) in accordance with current data protection regulations.

Statistical analysis All study variables were examined to assess their distribution. Categorical variables were described using the percentage associated with each possible response option, and quantitative variables using the mean, standard deviation (SD), and range. For comparisons between variables and the hypothesis test, the chi-square test was used for categorical variables, Student's t-test or ANOVA for quantitative variables that were normally distributed, and the Mann-Whitney U test or Kruskal-Wallis test for quantitative variables without normal distribution. Statistical analysis was performed with the SPSS v26 package (IBM, Armonk, New York).

ELIGIBILITY:
Inclusion criteria:

* Students over 18 years of age
* Students enrolled in the second year of the Bachelor's Degree in Nursing
* Students belonging to the Complutense University of Madrid

Exclusion criteria:

* Some physical inability to perform the impedance
* Failure to take exams
* Taking pharmacological treatments such as thyroid hormones, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: students of the Faculty of Nursing of the Complutense University of Madrid
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
KIDMED Questionnaire | 6 months
  This questionnaire will be taken by the students before and after the exam period to see if the score obtained from it varies
  Quiz Score:
  KIDMED Index Value
  ≤ 3: Very low-quality diet 4 to 7: Need to improve the dietary pattern to adjust it to the Mediterranean model.
  * 8: Optimal Mediterranean diet
  The sums of the positive values were classified into three levels:
  * 8-12: Optimal Mediterranean diet (high adherence)
  * 4-7 improvement needed to adjust intake to Mediterranean patterns (medium adherence)
  * 0-3 very low diet quality (low adherence)
INTERNATIONAL PHYSICAL ACTIVITY QUESTIONNAIRE (IPAQ) | 6 months
  This questionnaire will be taken by the students before and after the exam period to assess if there are changes in the score
  Value of the test:
  * Vigorous physical activity: 8 METs X minutes x days per week
  * Moderate physical activity: 4 METs x minutes x days per week
  * Walking: 3.3 x minutes x days per week EXAMPLE: 8 MET X 30 minutes x 5 days = 1200 MET (INTENSE PHYSICAL ACTIVITY)
  Next, add up the three values obtained:
  TOTAL: Vigorous physical activity + moderate physical activity + walking
Fat mass | 6 months
  Fat mass will be measured with a bioimpedance meter before and after the examination period to assess whether there are variations in the results obtained
Muscle mass | 6 months
  Muscle mass will be measured with a bioimpedance meter before and after the examination period to assess whether there are variations in the results obtained
Visceral tissue | 6 months
  Visceral tissue will be measured with a bioimpedance meter before and after the examination period to assess whether there are variations in the results obtained

SECONDARY OUTCOMES:
Age | 6 months
  Write down the student's age
Smoker | 6 months
  Write down whether or not the student smokes before and after the exam period
caffeine or cola drinks | 6 months
  The student will be asked if they drink caffeine or cola drinks before and after the exams
Height | 6 months
  Height will be measured with a bioimpedance meter before and after the examination period to assess whether there are variations in the results obtained
Weight | 6 months
  Weight will be measured with a bioimpedance meter before and after the examination period to assess whether there are variations in the results obtained
Body mass index (BMI) | 6 months
  BMI will be measured with a bioimpedance meter before and after the examination period to assess whether there are variations in the results obtained

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Publication of the study
Supporting Information: Study Protocol
Time Frame: Finals 2025